CLINICAL TRIAL: NCT01557946
Title: Glutamatergic and GABAergic Mediators of Antidepressant Response in Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Brian P. Brennan, MD, Associate Director of Translational Neuroscience Research, Mclean Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-P-001192
Record Dates: First submitted 2012-03-09; First posted 2012-03-20 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: MDD; Citalopram; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Citalopram

STUDY DESIGN:
Intervention Model Description: Open-label administration of citalopram to participants with major depressive disorder. MRI scans performed at baseline and days 3, 7, and 42. An age- and gender-matched group of healthy volunteers did not receive citalopram and received on MRI scan to perform between-group baseline analyses.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Major Depression (Experimental): Participants with major depressive disorder received citalopram 20-40 mg daily for 6 weeks. MRI scans were acquired at baseline and days 3, 7, and 42.
  Interventions: Drug: citalopram
- Healthy Volunteers (No Intervention): Healthy volunteer participants did not receive citalopram and performed one MRI scan.

INTERVENTIONS:
Drug: citalopram — citalopram 20-40 mg daily
  Other Names: Celexa
  Arms: Major Depression

SUMMARY:
Primarily, this study seeks to evaluate whether citalopram treatment is associated with an increase in the Glutamine (Gln)/Glutamate (Glu) ratio in the anterior cingulate cortex (ACC) from baseline to day 3 of treatment. Additionally, this study would like to examine whether citalopram treatment is associated with an increase in the Gln/Glu ratio in the ACC from baseline to day 7 of treatment. In order to more fully examine baseline neurochemical and functional abnormalities in participants with MDD, we also seek to scan a group of age- and sex-matched non-depressed comparison individuals in order to perform between-group analyses of baseline neuroimaging measures.

DETAILED DESCRIPTION:
Little is known about the acute effects of standard antidepressant treatments on brain glutamate and gamma-amino-butyric acid (GABA) levels, and their association with clinical response. In the current study, we used proton magnetic resonance spectroscopy (1H-MRS) to examine longitudinally the effects of citalopram on the glutamine/glutamate ratio and GABA levels in the pregenual anterior cingulate cortex (pgACC) - a region that has been repeatedly implicated in antidepressant response - of individuals with major depressive disorder (MDD). We acquired 1H-MRS scans at baseline and at days 3, 7, and 42 of citalopram treatment in nineteen unmedicated individuals with MDD. Ten age- and sex-matched non-depressed comparison individuals were scanned once and did not receive citalopram. The association between baseline metabolites and the change in metabolites from baseline to each time point and change in Montgomery-Åsberg Depression Rating Scale (MADRS) score from baseline to day 42 was assessed by longitudinal regression analysis, adjusting for age, sex, and baseline MADRS, using generalized estimating equations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 18 and ≤ 65
2. Meets DSM-IV criteria for MDD
3. Current score of ≥ 18 on the 21-item Hamilton Depression Rating Scale (HAM-D).

Exclusion Criteria:

1. Unwillingness or inability to provide written informed consent.
2. Current suicidal ideation
3. Active psychotic symptoms
4. Lifetime history of bipolar disorder, schizophrenia, or OCD
5. Failed treatment with an adequate trial of ≥ 2 antidepressants during the current major depressive episode ("failure" will be defined as ≤ 50% subjective improvement, and an "adequate trial" will be defined as at least 4 weeks of treatment using at least the minimum dose of the antidepressant recommended by the manufacturer in product labeling)
6. DSM-IV diagnosis of alcohol or substance dependence, with the exception of nicotine dependence, within three months prior to screening
7. Any history of treatment with electroconvulsive therapy
8. Positive urine toxicology screen for any drug of abuse or excluded medication at screening. Opiate pain medication being taken for a medical condition is exempt from needing a negative opiate screen.
9. Clinically significant medical or neurologic disease, as judged by the principal investigator, which would increase the risk to the participant or interfere with interpretation of results
10. Female participants with a positive urine pregnancy test at screening

12. Pregnancy. Females of childbearing potential must be using an effective contraceptive method (e.g., abstinence, prescription oral contraceptives, contraceptive injections, double-barrier method, male partner sterilization).

13. Any screening laboratory abnormality deemed clinically significant by the investigator 14. A QTc interval on screening ECG of ≥ 450 msec. 15. Use of any excluded medications (see Section 6.7 below) that cannot be discontinued during the screening phase 16. Previous failure to respond to treatment with citalopram that would, in the judgment of the investigator, constitute an adequate trial in MDD 17. Treatment with any investigational medications within 30 days prior to screening 18. Any contraindications to having an MRI scan, including cardiac pacemakers, metal vascular clips or stents, artificial heart valves, certain kinds of prostheses, brain stimulator devices, implanted drug pumps, ear implants, eye implants or known metal fragments in eyes, exposure to shrapnel or metal filings (wounded in military combat, sheetmetal workers, welders, and others), transdermal drug delivery systems, and certain tattoos with metallic ink 19. Left-handedness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P. Brennan, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Citalopram 20 mg / 40 mg: Citalopram tablet taken once daily.
  Only applicable to MDD participants. Every subject began on 20 mg, and had the option to titrate up to 40 mg.
- Healthy Control: No citalopram tablet taken.
Period: Overall Study
Arm/Group | Citalopram 20 mg / 40 mg | Healthy Control
Started | 20 | 12
Completed | 17 (20 consented and scanned - 1 subject's data not used due to ongoing neurological condition.) | 12 (2 subjects with unusable imaging data.)
Not Completed | 3 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Citalopram 20/40 mg: Citalopram tablet taken once daily.
- Total: Total of all reporting groups
Arm/Group | Citalopram 20/40 mg | Healthy Control | Total
Number analyzed (Participants) | 20 | 12 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 12 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.7) | 38.2 (14.1) | 39.0 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 12 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 16 | 7 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference From Baseline to Day 3 in Glutamine/Glutamate (Gln/Glu) Ratio Within Depressed Group
Description: Estimated mean difference (day 3 minus baseline) in the glutamine/glutamate (Gln/Glu) ratio in the rostral anterior cingulate cortex as measured by proton magnetic resonance spectroscopy from baseline to day 3 of citalopram treatment within the depressed group. The change in metabolites from baseline to each time point was assessed by random regression analysis, adjusting for age and sex, using generalized estimating equations to account for the correlation of observations within individuals.
Time Frame: Change from Baseline to Day 3
Population: One participant lacked a day 3 scan; one participant's day 3 scan was corrupted during data transfer and could not be recovered; and one participant's day 3 scan data was judged to be unusable due to poor spectral quality. Results are only presented for participants with depression as healthy control participants were only scanned once.
Measure: Mean (Standard Error); unit: arbitrary units
Groups:
- Participants With Depression: Participants with depression receiving citalopram
Arm/Group | Participants With Depression
Number analyzed (Participants) | 16
arbitrary units | 0.015 (0.032)

2. Secondary Outcome: Mean Difference From Baseline to Day 7 in Glutamine/Glutamate (Gln/Glu) Ratio Within Depressed Group
Description: Estimated mean difference (day 7 minus baseline) in the glutamine/glutamate (Gln/Glu) ratio in the rostral anterior cingulate cortex as measured by proton magnetic resonance spectroscopy from baseline to day 7 of citalopram treatment within the depressed group. The change in metabolites from baseline to each time point was assessed by random regression analysis, adjusting for age and sex, using generalized estimating equations to account for the correlation of observations within individuals.
Time Frame: Change from baseline to day 7
Population: One participant's day 7 scan was corrupted during data transfer and could not be recovered. Results are only presented for participants with depression as healthy control participants were only scanned once.
Measure: Mean (Standard Error); unit: arbitrary units
Arm/Group | Participants With Depression
Number analyzed (Participants) | 18
arbitrary units | -0.0025 (0.031)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the duration of participant's participation in study (on average 8 weeks). Adverse events relate specifically to study medication.
Groups:
- Citalopram 20 mg / 40 mg: Citalopram tablet taken once daily.
Arm/Group | Citalopram 20 mg / 40 mg | Healthy Control
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/0
Other Adverse Events (participants affected / at risk) | 19/19 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Citalopram 20 mg / 40 mg (N=19) | Healthy Control (N=0)
Headaches (General disorders) | 9 | 0
Insomnia (General disorders) | 6 | 0
Nausea (General disorders) | 4 | 0
Sedation (General disorders) | 4 | 0
Teeth Grinding (General disorders) | 3 | 0
Vivid Dreams (General disorders) | 2 | 0
Lethargy (General disorders) | 3 | 0
"Emotional Dulling" (Psychiatric disorders) | 1 | 0
Abdominal Cramping (Gastrointestinal disorders) | 1 | 0
Anorgasmia (Reproductive system and breast disorders) | 2 | 0
Dry Mouth (General disorders) | 2 | 0
Increased Sweating (General disorders) | 2 | 0
Jaw clenching (General disorders) | 1 | 0
Lightheadedness (General disorders) | 1 | 0
Decreased Libido (Reproductive system and breast disorders) | 1 | 0
"Heaviness in Eyelids" (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
"Spaciness" (General disorders) | 1 | 0
Dizziness (General disorders) | 1 | 0
Palpitations (General disorders) | 1 | 0
Right-Sided Jaw Pain (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Modest sample size due to participant attrition and the cost and logistical challenges of the study design.

Multiple comparisons, increasing the likelihood of type I errors. Open-label design which leaves open the possibility of a placebo effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No